CLINICAL TRIAL: NCT04342078
Title: Vitamin D and Health Outcomes in Preterm Born Population -A Cohort and an Intervention Study of Vitamin D on Health Outcomes of Bones, Teeth, Muscles, Heart, and Lungs in Children and Adults Born Preterm in Northern Finland
Brief Title: Vitamin D and Health Outcomes in Preterm Born Population
Acronym: ViDePrePop
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: EETTMK 92/2017
Record Dates: First submitted 2019-05-16; First posted 2020-04-10 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-10

CONDITIONS: Vitamin D3 Deficiency; Prematurity; Lung Diseases; Heart Rate Variability; Stress Physiology; Bone Diseases, Metabolic
Keywords: Vitamin D; Prematurity; Bone mineralisation; Lung function; Heart rate; DXA
MeSH Terms: conditions — Premature Birth; Lung Diseases; Bone Diseases, Metabolic | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preterm Child group: Preterm children at the age of 5 years; Born before 34 gestation weeks in 2014-2017; Cared in Oulu University Hospital
- Preterm Adult group: Preterm born adults at the age of 24-25 years; Born before 34 gestation weeks in 1994-1997; Cared in Oulu University Hospital
  Interventions: Dietary Supplement: Vitamin D
- Adult Control group: Age and gender matched term born controls for comparison of the entry assessments in the Preterm Adult group

INTERVENTIONS:
Dietary Supplement: Vitamin D — To investigate the effect of one year vitamin D supplementation in preterm born adults (4000 IU = 100 micrograms a day if serum concentration is < 30 nmol/l, 2000 IU = 50 micrograms a day if 30-50 nmol/l and 1000 IU = 25 micrograms a day if > 50-80 nmol/l, and no additional supplement if > 80 nmol/l) on health outcomes (bones, teeth, muscles, heart, lungs) . The target level of vitamin D concentration by every 4 months interval is 80 - 120 nmol/l .(Preterm Adult group)
  Groups: Preterm Adult group

SUMMARY:
Improved survival of very preterm newborn population during the last decades has challenged us neonatologists to study and improve nutritional practices including vitamin D (VitD) supplementation. However, long term outcome in this aspect has not been researched in well documented preterm populations. As VitD has receptors in almost all human cells it modulates growth of many organs. Therefore I start to assess VitD supplementation practices and later health outcome (bones, teeth, muscles, heart, lungs) in two preterm population cohorts cared in Oulu University Hospital at the age of 5 years and 24 years (born 2014-2017 and 1994-1997).

DETAILED DESCRIPTION:
Goals:

* To investigate the impact of VitD and mineral supplementation and biochemistry in infancy on health outcomes at the age of 5 years in childhood (bones, teeth, muscles, heart, lungs) after preterm birth (Preterm Child group)
* To investigate the impact of VitD and mineral supplementation and biochemistry in infancy on health outcomes at the age of 24-25 years in adulthood (bones, teeth, muscles, heart, lungs) after preterm birth (Preterm Adult group)

Subjects:

* Preterm Child group; Children, who were born prematurely before before 32 gestation weeks and before 34 gestation weeks with very low birth weight (VLBW, < 1500g) in Oulu University Hospital and/or cared in Neonatal Unit with VitD concentration measured before discharge during the years 2014 to 2017.
* Preterm Adult group; Adults, who were born prematurely before 32 gestation weeks and before 34 gestation weeks with very low birth weight (VLBW, < 1500g) in Oulu University Hospital and/or cared in Neonatal Intensive Unit during the years 1994 to 1997. For power calculation, the amount of participants for the adult group was done by estimating the inadequately low vitamin D concentration (< 50 nmol/l) to be found in 28 % of preterm born adults. (In Northern Finnish birth cohort 28 % at the age of 31 had serum 25-OH vitamin D concentration < 50 nmol/l in 1997). With the estimation of supplementation to decrease the percentage of participants with low vitamin D to 9 %, the required amount of participants would be minimum of 56 per group. Furthermore, if the level after supplementation is estimated to be low only in 2,8 %, the amount would be required as 29 cases per group.

Methods in protocol:

At the first visit and in the end of intervention; measurements of length, weight, head circumference, waist-to-hip ratio will be done; muscular power is assessed by grip test of both hands; lung function test with bronchodilatation is done at the first appointment; heart ultrasound, blood pressure measurement and bicycle stress test with a circadian electrocardiography will be done in the beginning and at the end; bone mineralisation will be measured by dual energy x-ray absorptiometry (DXA) and ultrasound methods; VitD concentration will be measured 4 months interval during the follow up. The control peers participate only the first visit. The child group will be assessed only once and without bicycle stress test.

ELIGIBILITY:
Inclusion Criteria:

* preterm and term born adults at the age of 22-25
* preterm born children at 5 years

Exclusion Criteria:

- motor disability

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy preterm born children and young adults. Tern born young adults as controls for the adult group.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin D of preterm adults, before = VitD 0A | Baseline
  S-25-OH -value; nmol/l
Vitamin D of preterm children = VitD C | Baseline
  S-25-OH -value;nmol/l
Vitamin D of preterm adults, after = VitD 1A | One year
  S-25-OH -value; nmol/l
Exercise heart rate, before = HR 0A | Baseline
  Cycling stress test; heart rate following maximal exercise , seconds to hours
Exercise heart rate, after = HR 1A | One year
  Cycling stress test;heart rate following maximal exercise , seconds to hours
HRV of preterm adults, before = HRV 0A | Baseline
  Heart rate variability; autonomic function; heart rate root mean square of the successive differences (RMSSD)
HRV of preterm adults, after = HRV 1A | One year
  Heart rate variability; autonomic function; heart rate root mean square of the successive differences (RMSSD)
HRV of preterm children = HRV 0C | Baseline
  Heart rate variability; autonomic function; heart rate root mean square of the successive differences (RMSSD)
Lung reversibility test in preterm adults, before = LR 0 | Baseline
  Spirometry and bronchodilate test; reversibility: Yes or No
Lung function capacity in preterm adults, before = LFC 0 | Baseline
  Spirometry; z-score of FVC
Lung function volume in preterm adults, before = LFV 0 | Baseline
  Spirometry ; z-score of FEV1
Lung function capacity in preterm adults, after = LFC 1 | One year
  Spirometry; z-score of FVC
Lung function volume in preterm adults, after = LFV 1 | One year
  Spirometry; z-score of FEV1
Lung function in preterm children | Baseline
  Auscultation and bronchodilate test; reversibility: Yes or No
Body composition of bone mineral density in preterm adults, before = BMD 0A | Baseline
  DXA result; bone mineral density (BMD) g/cm2; Z-scores
Body composition of bone mineral content in preterm adults, before = BMC 0A | Baseline
  DXA result; bone mineral content (BMC) g; Z-scores
Body composition of bone mineral density in preterm children = BMD C | Baseline
  DXA result; bone mineral density (BMD) g/cm2; Z-scores
Body composition of bone mineral content in preterm children = BMC C | Baseline
  DXA result; bone mineral content (BMC) g; Z-scores
Body composition of bone mineral density in preterm adults, after = BMD 1A | One year
  DXA result; bone mineral density (BMD) g/cm2; Z-scores
Body composition of bone mineral content in preterm adults, after = BMC 1A | One year
  DXA result; bone mineral content (BMC) g Z-scores

OTHER OUTCOMES:
Bone mineralisation, before = BM 0 | Baseline
  ultrasound; bone speed of sound (SOS) m/sec z-score
Bone mineralisation, after = BM 1 | One year
  ultrasound; bone speed of sound (SOS) m/sec z-score

CONTACTS AND LOCATIONS:
Overall Officials: Marita Valkama, Docent, Study Chair — MRC, University of OUlu; Marja Ojaniemi, Docent, Study Director — MRC, University of Oulu
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No